CLINICAL TRIAL: NCT05553652
Title: The Effect of ASTARTE™; Lactobacillus Crispatus, Lactobacillus Rhamnosus, Lactobacillus Jenesii and Lactobacillus Gasseri on the Reduction of Risk Factors for Recurrent Urinary Tract Infection in Women
Brief Title: The Effect of ASTARTE™ on Recurrent Urinary Tract Infection
Acronym: rUTI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Andreas Munk Petersen, MD, Associate Professor, PhD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: H-22014666
Record Dates: First submitted 2022-09-16; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Recurrent Urinary Tract Infection
Keywords: rUTI; Probiotic
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASTARTE™ oral capsule (Active Comparator): The capsule will contain a mixture of four probiotic strains with a combined potency of 5 x10^9 (CFU)/capsule:
  Lactobacillus crispatus LBV88, 2 x10^9 CFU/g Lactobacillus rhamnosus LBV96, 2 x10^9 CFU/g Lactobacillus gasseri LBV150N , 0.6 x10^9 CFU/g Lactobacillus jensenii LBV116, 0.4 x10^9 CFU/g Corn starch 79 mg, Magnesium salts of fatty acid 3 mg, Silicon dioxide 3 mg, Vegetal capsule size 1 DR white 75 mg, Fructooligosaccharides 30mg
  Interventions: Dietary Supplement: ASTARTE™ oral capsules; Dietary Supplement: Placebo oral capsules
- Placebo oral capsule (Placebo Comparator): The placebo oral capsules is identical to the ASTARTE™ capsules and contains Corn starch 79 mg, Magnesium salts of fatty acid 3 mg, Silicon dioxide 3 mg, Vegetal capsule size 1 DR white 75 mg, Fructooligosaccharides 30mg
  Interventions: Dietary Supplement: ASTARTE™ oral capsules; Dietary Supplement: Placebo oral capsules

INTERVENTIONS:
Dietary Supplement: ASTARTE™ oral capsules — 1 Capsule daily for 6 months
Dietary Supplement: Placebo oral capsules — 1 Capsule daily for 6 months

SUMMARY:
Investigate the effect of dietary supplements/probiotic ASTARTE™ ( L. crispatus, L. rhamnosus, L. jensenii, L. gasseri) on the microbiome composition in the intestine and vagina and thereby a reduction of risk factors for the development of rUTI during 6 months of intervention in women aged 18-40 years. This is measured by the incidence of symptomatic UTI.

DETAILED DESCRIPTION:
Urinary tract infection (UTI) is one of the most common infections, contributing to increased antibiotic consumption and high costs. Women are often developing UTI due to the anatomically short distance from the rectum opening to the urethra. There is a risk of serious complications associated with pregnancy, where there is an increased risk of developing pelvic inflammatory disease and premature birth. This will in some cases lead to increased risk of maternal and neonatal morbidity and mortality; especially in infection with Streptococcus agalactiae. Recurrent UTI (rUTI) with urease producing microorganisms such as Proteus and Klebsiella will cause an increased risk of developing stones in the urinary tract.

Scientific studies suggest that probiotics can be effective dietary supplements reducing the risk factors for the development of infections in the intestine and vagina. Probiotics are non-pathogenic microorganisms capable of affecting gastrointestinal microbiota with a change in microbiota composition, thus increasing the production of beneficial substances when ingested in appropriate quantities. The consumption of probiotics is not considered to be associated with adverse reactions to humans because they are usually found naturally in e.g. gastrointestinal and vaginal microbiota.

A prospective study over 2-years which is conducted as a randomized placebo-controlled double-blind study. In this study the investigators will investigate the effect of probiotics ASTARTE™ ( Lactobacillus crispatus, Lactobacillus rhamnosus, Lactobacillus jensenii, Lactobacillus gasseri) on the composition of bacteria in urine, faces and vagina, and a possible reduction of risk factors for development of rUTI in women (18 to 40 years). The investigators will map the microbiota in the faeces and vagina and examine if there are a relationship between colonization of the urinary tract with pathogens and the composition of the intestinal and vaginal microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-40 years of age
* Recurrent UTI (2 times UTI within 6 months or > 3 times UTI infection within one year).
* The subjects should be informed about the trial protocol.
* The subject must be able to follow the protocol, have provided voluntary consent and have signed the declaration of consent.

Exclusion Criteria:

* Pregnancy or planning pregnancy
* Breastfeeding
* Participation in another trial with probiotic the last 30 days.
* Hypersensitivity to any ingredient in the study product
* Patients primarily admitted for a disorder other than UTI
* Antibiotic treatment for any other condition than UTI at time of recruitment the last 30 days

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women 18-40 years of age, Recurrent UTI (2 times UTI within 6 months or > 3 times UTI infection within one year).
Enrollment: 720 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of UTI cases | 6 months
  Number of symptomatic urinary tract infection cases during the intervention compared to the number of UTI cases before the intervention (> 2 UTIs per year). Measured from a urine sample.

SECONDARY OUTCOMES:
Number of UTI after intervention | 12 months
  Number of symptomatic urinary tract infection cases during the intervention compared to the number of UTI cases after the intervention. Measured from a urine sample.
UTI symptoms | 12 months
  Change in UTI symptoms from the baseline measure by the ICIQ-FLUTS questionnaire every 2d months. We measure score values:
  0-16 filling symptoms subscale, 0-12 voiding symptoms subscale, 0-20 incontinence symptoms subscale
Change of vaginal microbiome | 6 months
  Change in vaginal microbiome from the baseline measure by Microbiome genetic test. Measure from a feacal sample every 2d month in the intervention period.
Change of gut microbiome | 6 months
  Change in gut microbiome from the baseline measure by Microbiome genetic test. Measure from a fecal sample every 2d month in the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Petersen, DM. PhD, Principal Investigator — Hvidovre Hospital, University of Copenhagen
Locations (1):
- Gastrounit, Copenhagen University Hospital Hvidovre, Hvidovre, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No